CLINICAL TRIAL: NCT00873119
Title: An Open-label Randomized Phase II Trial of Belinostat (PXD101) in Combination With Carboplatin and Paclitaxel (BelCaP) Compared to Carboplatin and Paclitaxel in Patients With Previously Untreated Carcinoma of Unknown Primary
Brief Title: Belinostat, Carboplatin and Paclitaxel (BelCaP) Compared to Carboplatin and Paclitaxel in Patients With Cancer of Unknown Primary
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valerio Therapeutics (Industry)
Collaborators: Spectrum Pharmaceuticals, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PXD101-CLN-17
Record Dates: First submitted 2009-03-31; First posted 2009-04-01 (Estimated); Results first posted 2014-12-09 (Estimated); Last update posted 2015-07-28 (Estimated); Status verified 2015-07

CONDITIONS: Carcinoma of Unknown Primary
Keywords: Belinostat; PXD101; Carboplatin; Paclitaxel; CUP; Carcinoma of unknown primary; Occult primary
MeSH Terms: conditions — Neoplasms, Unknown Primary | interventions — belinostat; Carboplatin; Paclitaxel; CP protocol

ARMS (2):
- Arm A - BelCaP (Experimental): Group A: belinostat 1000 mg/m² administered as a 30 minute IV infusion once daily on days 1, 2 and 3, with at least 18 hours between infusions, followed by belinostat 2000 mg administered orally once daily on days 4 and 5, every 3-weeks, in combination with paclitaxel 175 mg/m² administered as an IV infusion following the infusion of belinostat on cycle day 3, and carboplatin (AUC 6) administered as a 30-60 minute IV infusion directly after the paclitaxel administration on cycle day 3.
  Interventions: Drug: belinostat, carboplatin, paclitaxel
- Arm B - CaP (Active Comparator): Group B: paclitaxel 175 mg/m² administered as an IV infusion directly followed by carboplatin (AUC 6) administered as a 30-60 minute IV infusion on cycle day 1 of a 3-weekly cycle.
  Interventions: Drug: carboplatin, paclitaxel

INTERVENTIONS:
Drug: belinostat, carboplatin, paclitaxel
  Other Names: PXD101, Belinostat; Carboplatin; Paclitaxel, Taxol
  Arms: Arm A - BelCaP
Drug: carboplatin, paclitaxel
  Other Names: Carboplatin; Paclitaxel, Taxol
  Arms: Arm B - CaP

SUMMARY:
The purpose of this study is to assess efficacy and safety of belinostat in combination with carboplatin and paclitaxel in patients with previously untreated carcinoma of unknown primary.

DETAILED DESCRIPTION:
This is an open-label, multinational, multicenter, randomized, comparative efficacy and safety study in previously untreated patients with carcinoma of unknown primary. Patients meeting inclusion and exclusion criteria will be randomized to treatment in Arm A (BelCaP) or Arm B (CaP).

ELIGIBILITY:
Inclusion Criteria:

* Patients with CUP where the primary site had not been revealed by complete history, physical examination (including gynecological examination when appropriate), computed tomography (CT) scan of the chest, abdomen and pelvis, bilateral mammography (in women with adenocarcinoma or poorly differentiated carcinoma), routine laboratory studies (complete blood cell counts, electrolytes, urinalysis, liver and renal function tests), and directed work-up of any other symptomatic areas.
* Light microscopic pathologic diagnosis of adenocarcinoma (including poorly differentiated), squamous cell carcinoma, or poorly differentiated carcinoma. Patients with poorly differentiated carcinoma must have immunohistochemical stains to confirm the diagnosis of carcinoma, and to rule out other tumor types. Note: patients with a light microscopic histology diagnosis of "poorly differentiated neoplasm, not otherwise classified" did not fulfill the criteria for inclusion, unless immunohistochemical staining confirmed the diagnosis of carcinoma.
* Signed consent of an IRB ([Institutional Review Board])/IEC ([Independent ethics committee]) approved ICF ([Informed Consent Form]).
* At least one measurable lesion according to RECIST ([response evaluation criteria in solid tumors ]) criteria. Note, target lesions could only be selected within previously irradiated areas if newly arising or clearly progressing after irradiation as proven by repeat scanning
* Performance status Eastern Cooperative Oncology Group (ECOG) ≤ 2.
* Age ≥ 18 years.
* A negative serum or urine pregnancy test for women of childbearing potential. Postmenopausal women must have been amenorrheic for ≥ 12 months to be considered of non-childbearing potential.
* Serum potassium within normal range.
* Acceptable coagulation status: Prothrombin time/International normalized ratio PT/INR ([international normalized ratio]), and activated partial thromboplastin time (APTT) ≤ 1.5 × upper limit of normal (ULN) or in the therapeutic range if on anticoagulation therapy.
* Acceptable liver, renal and bone marrow function including the following:

  1. Bilirubin ≤ 1.5 times ULN (if liver metastases were present, then ≤ 3 × ULN was allowed).
  2. Aspartate aminotransferase/serum glutamic oxaloacetic transaminase (AST/SGOT), alanine amino transferase/serum glutamic pyruvic transaminase (ALT/SGPT), and alkaline phosphatase ≤ 3 times ULN (if liver metastases were present, then ≤ 5 × ULN was allowed).
  3. An estimated creatinine clearance ≥ 45 mL/min using an appropriate formula (Appendix C, protocol version 1.0, Appendix 16.1.1), or measured ethylenediaminetetraacetic acid (EDTA) renal clearance ≥ 45 mL/min.
  4. Absolute neutrophils count ≥ 1.5 × 109/L, platelets ≥ 100 × 109/L.
  5. Hemoglobin ≥ 9.0 g/dL or ≥ 5.6 mmol/L (patients with chronic anemia due to underlying disease and its treatment could undergo blood transfusion prior to treatment in order to meet this criteria).

Exclusion Criteria:

* Patients with well recognized subsets of CUP site where treatments directed towards a defined tumor type, or surgery, alternatively radiotherapy, can be advised:
* Women with adenocarcinoma involving only axillary lymph nodes.
* Women with papillary serous carcinoma of the peritoneum.
* Women with adenocarcinoma with positive staining for estrogen receptor (ER) or progesterone receptor.
* Young men (< 45 years) with poorly differentiated carcinoma consistent with an extragonadal germ cell tumor (carcinoma involving mediastinum or retroperitoneum, or elevated levels of beta-human chorionic gonadotropin or alpha-fetoprotein).
* Men with bone metastases and/or adenocarcinoma, and abnormally elevated PSA ([Prostate specific antigen]) in their plasma.
* Patients with squamous cell carcinoma involving only cervical lymph nodes, or inguinal lymph nodes.
* Patients with neuroendocrine carcinomas determined according to standard pathology diagnosis procedures, including stains.
* Patients with potentially completely resectable metastatic disease, or disease which can be adequately treated with radiotherapy only.
* Patients with brain or meningeal metastases. Note, patients with adequately treated brain metastases, e.g. surgically resected, or adequately controlled by radiotherapy, with no residual neurological symptoms due to metastases and no steroid treatment required, could be enrolled. If clinical suspicion, adequate investigations should be performed to rule out brain metastases or meningeal involvement.
* Prior systemic anti-tumor therapy, including chemotherapy administered in association to radiotherapy for sensitization, for CUP. Note, prior radiotherapy or surgery was allowed provided treatment was completed at least 4 weeks before randomization.
* Treatment with investigational agents, including non-anti-tumor agents, within the last 4 weeks before randomization.
* Co-existing active severe infection or any co-existing medical condition assessed by the Investigator as likely to interfere with study procedures.
* Significant cardiovascular disease (New York Heart Association Class III or IV cardiac disease), myocardial infarction within the past 6 months, unstable angina, unstable arrhythmia or a need for anti-arrhythmic therapy (use of medication to control heart rate in patients with atrial fibrillation was allowed, if on stable medication for at least the last month prior to randomization and the medication not listed as causing Torsade de Points (Section 13.2, Appendix B, protocol version 1.0, Appendix 16.1.1), or evidence of acute ischemia on ECG.
* Marked baseline prolongation of QT/QTc ([corrected QT interval]) interval, i.e., demonstration of a QTc interval > 450 millisecond (ms); Long QT Syndrome; the required use of concomitant medication that may cause Torsade de Pointes (Section 13.2, Appendix B, protocol version 1.0, Appendix 16.1.1).
* Altered mental status precluding understanding of the informed consent process and/or completion of the necessary study procedures.
* History of a previous malignancy within 5 years with the exception of non-metastatic non-melanoma skin cancer or cervical carcinoma in situ. Prior systemic therapy for other malignancy completed at least 5 years before randomization is allowed.

Implemented with amendment 2 (study centers in France only): History of a previous malignancy, irrespective of time since diagnosis/treatment, with the exception of non metastatic non-melanoma skin cancer or cervical carcinoma in situ.

* Known hypersensitivity to either platinum compounds or paclitaxel, or any components of the study medications, and inability for desensitization.
* Known infection with HIV, or known active Hepatitis B or C infection.
* Peripheral neuropathy ≥ Grade 2.
* Pregnant or lactating females.
* Women of childbearing age and potential who are not willing to use effective contraception during the study and until 30 days after last dose of study drug. Male patients or male patients who have female partners of childbearing age and potential who are not willing to use effective contraception during the study and until 30 days after last dose of study drug. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1% per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, some intra uterine devices, sexual abstinence or vasectomized partner.
* Patients that are not affiliated with social security (study centers in France only).
* Implemented with amendment 1 (study centers in Denmark only): Hearing impairment assessed by the Investigator as being of such a degree that treatment with carboplatin cannot be initiated.
* Implemented with amendment 1 (study centers in Denmark only): Bleeding tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2009-02; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: e-mail contact via enquires@topotarget.com, Study Director — Valerio Therapeutics
Locations (23):
- United States (11):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Northwest Georgia Oncology Centers, Marietta, Georgia
  - Baton Rouge Medical Center, Baton Rouge, Louisiana
  - Center for Cancers and Blood Disorders, Bethesda, Maryland
  - Research Medical Center, Kansas City, Missouri
  - Oncology Hematology Care Inc., Cincinnati, Ohio
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Chattanooga Oncology & Hematology Associates, PC, Chattanooga, Tennessee
  - Tennessee Oncology Sarah Cannon Research, Nashville, Tennessee
  - South Texas Oncology and Hematology, San Antonio, Texas
  - Virginia Cancer Institute, Richmond, Virginia
- H:S Rigshospital, The Finsen Centre, Copenhagen, Denmark
- France (7):
  - CRLCC Francois Baclesse, Oncologie medicale, Caen
  - Centre Oscar Lambert, Lille
  - Centre Léon Bérard, Oncologie, Lyon
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Oncologie Médicale, Rouen
  - Institut de Cancerologie de la Loire, Saint-Priest-en-Jarez
  - Institut Gustave Roussy IGR, Villejuif
- Germany (4):
  - Carl-Gustav-Carus Medicinische Klinik und Poliklinik I, Dresden
  - Kliniken Essen-Mitte, Essen
  - ASKLEPIOS Klinik Altona, Hamburg
  - Ostholstein-Onkologie, Oldenburg in Holstein

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A - BelCaP: Group A: belinostat (1000 mg/m²) administered as a 30 minute IV infusion once daily on days 1, 2 and 3, with at least 18 hours between infusions, followed by belinostat (2000 mg) administered orally once daily on days 4 and 5, every 3-weeks, in combination with paclitaxel (175 mg/m²) administered as an IV infusion following the infusion of belinostat on cycle day 3, and carboplatin (AUC 6) administered as a 30-60 minute IV infusion directly after the paclitaxel administration on cycle day 3.
- Arm B - CaP: Group B: paclitaxel (175 mg/m²) administered as an IV infusion directly followed by carboplatin (AUC 6) administered as a 30-60 minute IV infusion on cycle day 1 of a 3-weekly cycle.
Period: Overall Study
Arm/Group | Arm A - BelCaP | Arm B - CaP
Started | 44 | 45
Completed | 0 (Of 42 patients treated with belinostat, 23 patients received 6 or more treatment cycles.) | 19
Not Completed | 44 | 26
Not completed — Patient request | 4 | 2
Not completed — Adverse Event | 8 | 0
Not completed — Progressive disease | 26 | 18
Not completed — Death | 2 | 1
Not completed — Other | 2 | 5
Not completed — Not treated | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - BelCaP | Arm B - CaP | Total
Number analyzed (Participants) | 44 | 45 | 89
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 31 | 60
  >=65 years | 15 | 14 | 29
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 23 | 47
  Male | 20 | 22 | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Time from the date of randomization to the time of disease progression or death due to any cause, measured by RECIST criteria (Response Evaluation Criteria In Solid Tumors).
Time Frame: Tumor assessment every 6 weeks for the treatment period. Subsequent assessments every 6 weeks for the initial 6 months, then every 9 weeks for 6 months, then every 12 weeks for 12 months and then every 6 months until 5 years from the start of study
Population: Intent-to-treat (ITT) population: All patients randomized to one of the two treatment groups were included in the ITT population, 12 patients (5 in Arm A and 7 in Arm B) were censored due to lack of efficacy
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - BelCaP | Arm B - CaP
Number analyzed (Participants) | 39 | 38
months | 5.4 [3.0 to 6.0] | 5.3 [2.8 to 6.7]

2. Secondary Outcome: Best Overall Response
Description: The best overall response in an individual patient according to the RECIST criteria (Eisenhauer 2009 ) is the best response recorded from the start of the treatment until disease progression/recurrence. Objective response is defined as best overall response of complete response (CR) or partial response (PR)
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population: All patients randomized to one of the two treatment groups were included in the ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Arm A - BelCaP | Arm B - CaP
Number analyzed (Participants) | 42 | 44
percentage of participants | 43.2 | 22.2

3. Secondary Outcome: Overall Survival (OS)
Description: Time from the date of randomization to the date of death
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population: All patients randomized to one of the two treatment groups were included in the ITT population. 18 patients (10 in Arm A and 8 in Arm B) were censored.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - BelCaP | Arm B - CaP
Number analyzed (Participants) | 34 | 37
months | 11.5 [6.9 to 18] | 9.1 [6.6 to 11]

4. Secondary Outcome: Time to Response
Description: For patients with overall best response being CR or PR, time to response was measured as the time from randomization to the first time when the measurement criteria for CR or PR (whichever status is recorded first) were met
Time Frame: as for outcome 1
Population: Patients with overall best response being either complete response or partial response.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A - BelCaP | Arm B - CaP
Number analyzed (Participants) | 19 | 10
months | 3.2 [0 to 19.1] | NA [0 to NA] — Median missing due to sparse data

5. Secondary Outcome: Duration of Response
Description: Duration of overall response was measured from the time that measurement criteria were first met for CR or PR (whichever status was recorded first) until the first date that PD ([Progressive Disease]) or death was documented
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population: All patients randomized to one of the two treatment groups were included in the ITT population. Three patients, 2 in Arm A and 1 in Arm B, were not treated with study medication
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - BelCaP | Arm B - CaP
Number analyzed (Participants) | 19 | 10
months | 4.6 [3.3 to 8.3] | 6.5 [2.9 to 24.2]

6. Secondary Outcome: Time to Progression (TTP)
Description: Time from the date of randomization to the time of disease progression
Time Frame: as for outcome 1
Population: Intent-to-treat (ITT) population: All patients randomized to one of the two treatment groups were included in the ITT population. 26 patients (12 in Arm A and 14 in Arm B) were censored. One patient in each arm had no information reported.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - BelCaP | Arm B - CaP
Number analyzed (Participants) | 31 | 30
months | 5.7 [4.5 to 7.2] | 5.6 [2.8 to 7.5]

ADVERSE EVENTS:
Description: Safety population consist of 86 of 89 included patients. 3 patients (2 in Arm A and 1 in Arm B) did not receive study medication
Arm/Group | Arm A - BelCaP | Arm B - CaP
Serious Adverse Events (participants affected / at risk) | 22/42 | 10/44
Other Adverse Events (participants affected / at risk) | 42/42 | 43/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - BelCaP (N=42) | Arm B - CaP (N=44)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 2
Hypersensitivity (Immune system disorders) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related infection (Infections and infestations) | 1 | 0
Retroperitoneal abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Panic attack (Psychiatric disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Arterial occlusive disease (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0
Venous stenosis (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Neutropenic infection (Infections and infestations) | 0 | 1
Pneunomia (Infections and infestations) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - BelCaP (N=42) | Arm B - CaP (N=44)
Nausea (Gastrointestinal disorders) | 36 | 26
Diarrhoea (Gastrointestinal disorders) | 24 | 17
Vomiting (Gastrointestinal disorders) | 26 | 13
Constipation (Gastrointestinal disorders) | 19 | 18
Abdominal pain (Gastrointestinal disorders) | 8 | 11
Dry mouth (Gastrointestinal disorders) | 6 | 1
Abdominal pain upper (Gastrointestinal disorders) | 4 | 2
Abdominal distension (Gastrointestinal disorders) | 3 | 2
Stomatitis (Gastrointestinal disorders) | 1 | 3
Fatigue (General disorders) | 27 | 29
Oedema peripheral (General disorders) | 10 | 10
Asthenia (General disorders) | 6 | 5
Pyrexia (General disorders) | 7 | 4
Chest pain (General disorders) | 5 | 2
Mucosal inflammation (General disorders) | 5 | 2
Chills (General disorders) | 3 | 2
Pain (General disorders) | 2 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 22 | 27
Rash (Skin and subcutaneous tissue disorders) | 10 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 14
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 11 | 6
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 3
Bone pain (Musculoskeletal and connective tissue disorders) | 3 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 5
Neuropathy peripheral (Nervous system disorders) | 15 | 8
Peripheral sensory neuropathy (Nervous system disorders) | 7 | 11
Dizziness (Nervous system disorders) | 6 | 7
Dysgeusia (Nervous system disorders) | 6 | 5
Headache (Nervous system disorders) | 5 | 6
Paraesthesia (Nervous system disorders) | 6 | 2
Decreased appetite (Metabolism and nutrition disorders) | 20 | 16
Dehydration (Metabolism and nutrition disorders) | 10 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 8
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 3
Anaemia (Blood and lymphatic system disorders) | 17 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 13 | 10
Neutropenia (Blood and lymphatic system disorders) | 14 | 8
Leukopenia (Blood and lymphatic system disorders) | 5 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 10
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 | 4
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 4
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Urinary tract infection (Infections and infestations) | 4 | 3
Nasopharyngitis (Infections and infestations) | 1 | 5
Oral candidiasis (Infections and infestations) | 3 | 1
Flushing (Vascular disorders) | 6 | 7
Hypotension (Vascular disorders) | 5 | 2
Phlebitis (Vascular disorders) | 3 | 1
Hot flush (Vascular disorders) | 0 | 3
Weight decreased (Investigations) | 4 | 5
Platelet count decreased (Investigations) | 3 | 4
Haemoglobin decreased (Investigations) | 3 | 2
Increased haemoglobin (Investigations) | 0 | 3
Neutrophil count decreased (Investigations) | 3 | 0
Insomnia (Psychiatric disorders) | 7 | 9
Anxiety (Psychiatric disorders) | 6 | 3
Drug hypersensitivity (Immune system disorders) | 6 | 5
Dysuria (Renal and urinary disorders) | 3 | 3
Tinnitus (Ear and labyrinth disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less